CLINICAL TRIAL: NCT01704118
Title: Is Size 1 I-gel More Effective Than Size 1 ProSeal Laryngeal Mask for Anesthetized Infants and Neonates?
Brief Title: Comparison of Size 1 I-gel and ProSeal Laryngeal Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gulay ERDOGAN KAYHAN, Assistant Prof,MD, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Inonu University
Record Dates: First submitted 2012-10-04; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Laryngeal Masks
Keywords: I-gel; ProSeal laryngeal mask; small infants; neonates

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I-gel (Experimental): I-gel (Intersurgical Ltd, Wokingham, Berkshire, UK) is a disposable supraglottic airway device with a non-inflatable cuff in which part of that is fixed on glottis is made of thermoplastic elastomer, unlike other laryngeal masks
  Interventions: Device: I-gel
- ProSeal Laryngeal mask (Active Comparator): ProSeal laryngeal mask (PLMA) (LMA North America, Inc., San Diego, USA) is a modified type of LMA (larger and deeper bowl and enlarged and softer cuff) with gastric drainage tube.
  Interventions: Device: ProSeal Laryngeal mask

INTERVENTIONS:
Device: I-gel — Supraglottic airway device
  Arms: I-gel
Device: ProSeal Laryngeal mask — Supraglottic airway device
  Other Names: PLMA
  Arms: ProSeal Laryngeal mask

SUMMARY:
Objective of this prospective, randomized and controlled study is to compare the performances of recently-released size 1 I-gel and size 1 PLMA proven to be superior to classical LMA with prospective studies. In this study, primer endpoint was value of airway leak pressure and secondary insertion time, insertion success and conditions, initial airway quality, hemodynamic parameters, fiberoptic view and complications will be assessed.

DETAILED DESCRIPTION:
Routine monitorization will be performed. Lidocaine 1 mg.kg-1, remifentanil 1 mcg.kg-1 (slow bolus in approximately 1 minute) and 3 mg.kg-1 propofol will be administered in anaesthesia induction.

In Group P, PLMA with fully deflated cuff and applied water-based lubricant, will be inserted using a metal introducer. After insertion, cuff will be inflated with a recommended volume of air and then cuff pressure will be adjusted to 60 cm H2O with manometer.

In Group I, I-gel with its cuff lubricated will be orally inserted along the hard palate until resistance will be felt, as recommended by the manufacturer.

The time between picking up the prepared PLMA (with introducer and deflated cuff) or I-gel and the appearance of the first stable capnographic trace will be recorded as the insertion time. The conditions for insertion will be ere scored according to mouth (1: full, 2: partial, 3: nil), gagging or coughing (1: nil, 2: slight, 3: gross), swallowing (1: nil, 2: slight, 3: gross), head or limb movement (1: nil, 2: slight, 3: gross), laryngospasm (1: nil, 2: slight, 3: complete) and ease of insertion (1: easy, 2: difficult, 3: impossible).

Fresh gas flow will be adjusted to 3 L.min-1, and after closing the expiratory valve the airway pressure at which an audible leak in the mouth occurred will recorded as the 'Pleak'. When Pleak reach 35 cm H2O, expiratory valve will be opened.

Anatomical position of airway device will viewed by inserting fiberoptic bronchoscope through the ventilation tube.

Complications encountered during and at the end of the operation such as desaturation (sPO2 less than 90%), gastric insufflation, aspiration, laryngospasm, bronchospasm and blood stain on the airway device during removal will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Infants and neonates, that to be used supraglottic airway and that plan to be taken elective surgery

Exclusion Criteria:

Infants having a history of pulmonary disease and expect to have aspiration (gastroesophageal reflux, gastrointestinal stenosis or stricture) and a difficult airway

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Airway leak pressure | 1 year (After anesthesia induction)
  Fresh gas flow will adjust to 3 L.min-1, and after closing the expiratory valve the airway pressure at which an audible leak in the mouth occurred will be recorded as the 'Pleak'.

SECONDARY OUTCOMES:
Insertion time and conditions | 1year (During maintainance of anesthesia)
  The time between picking up the device and the appearance of the first stable capnographic trace will be recorded as the insertion time. The conditions for insertion were scored according to mouth (1: full, 2: partial, 3: nil), gagging or coughing (1: nil, 2: slight, 3: gross), swallowing (1: nil, 2: slight, 3: gross), head or limb movement (1: nil, 2: slight, 3: gross), laryngospasm (1: nil, 2: slight, 3: complete) and ease of insertion (1: easy, 2: difficult, 3: impossible).
Initial airway quality | During maintainance of anesthesia
  Initial airway quality will be evaluated with manual ventilation by adjusting APL valve to 20 cm H2O. Evaluation will be performed with a scale as excellent (no leaks heard), good/acceptable (a slight, clinically insignificant leak, sufficient ventilation) and poor/unacceptable (significant leak and insufficient ventilation which requires reposition or relocation of device) by listening to lungs, epigastrium and perilaryngeal field and observing the expansion of thorax.
Evaluation of fiberoptic view | 1 year (During maintainance of anesthesia)
  The breathing system will be disconnected and fiberoptic bronchoscope will be inserted through the ventilation tube to evaluate glottic view. Fiberoptic images will be recorded by using a digital camera. The images will be graded according to the score of 1 to 5.
Complications | 1year(During maintainance of anesthesia)
  Complications encountered during and at the end of the operation such as desaturation, gastric insufflation, aspiration, laryngospasm, bronchospasm and blood stain on the airway device during removal will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gulay Erdogan Kayhan, Study Director — Assistant Professor, MD
Locations (1):
- Inonu University Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

REFERENCES:
- [Derived] Kayhan GE, Begec Z, Sanli M, Gedik E, Durmus M. Performance of size 1 I-gel compared with size 1 ProSeal laryngeal mask in anesthetized infants and neonates. ScientificWorldJournal. 2015;2015:426186. doi: 10.1155/2015/426186. Epub 2015 Feb 22. PMID 25793219